CLINICAL TRIAL: NCT01220830
Title: Efficacy of Rotational Field Quantum Nuclear Magnetic Resonance (RFQMR) Based Tissue Engineering in the Treatment of Multiple Sclerosis
Brief Title: Cytotron® Delivered Rotational Field Quantum Nuclear Magnetic Resonance Therapy for Multiple Sclerosis
Acronym: RFQMR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Centre for Advanced Research & Development, India (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100915_CIP_MS_V1.0
Record Dates: First submitted 2010-10-09; First posted 2010-10-14 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; RFQMR; Cytotron; EDSS; QOL assessment with FAMS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RFQMR on Multiple Sclerosis lesions (Experimental)
  Interventions: Device: Cytotron

INTERVENTIONS:
Device: Cytotron — Exposure to RFQMR with Cytotron for 28 consecutive days for one hour daily.
  Other Names: CYTOTRON-RTE-6040-844GEN

SUMMARY:
The purpose of the study is to evaluate the efficacy of RFQMR therapy in remyelination in cases of Multiple sclerosis.

The evaluation will be done based on MRI findings, by clinical/ neurological examination and by assessment of quality of life before and after completion of therapy.

DETAILED DESCRIPTION:
Transmembrane Potential (TMP) is one of the known cellular signalling pathways regulating synthesis of various proteins like those responsible for programmed cell death (e.g., p53 group) at the appropriate time in living cells. Many illnesses like cancer and degenerative diseases are linked to disturbances in transmembrane potential and protein transcription process.(Cone CD, 1970)

The protein responsible for production of myelin by the oligodendrocytes is Connexin 32. It has been established that in cases of Multiple Sclerosis (MS) this protein is not synthesized by the oligodendrocytes thus leading to non-repair of the demyelination process in the Central Nervous System (CNS) (Scherer SS et al., 1995; Sargiannidou I et al., 2009; Bondurand N et al., 2001). This causes the fibrotic damage and plaque formation and consequent signs and symptoms of MS. RFQMR therapy addresses this process of stimulation of Oligodendrocytes to synthesize Connexin 32 thus causing remyelination.

RFQMR therapy is delivered with CYTOTRON®. This device is a long body, wide bore machine with 864 guns, with near field antennae and parabolic reflector delivery system. The device is capable of producing a wide range of dosimetry, involving multiple modulations in both fixed and variable proton density dosimetry. Appropriately modulated multi-harmonic Radio Frequency (RF) signals in the lower end of the electromagnetic spectrum can be used in altering the cell signaling process using the TMP pathways, thus able to tackle systemic disorders. Generically known as Rotational Field Quantum Nuclear Magnetic Resonance (RFQMR), it is a technology that is made to deliver highly complex quantum instantaneous Nuclear Magnetic Resonance beams in the RF bands and its harmonics ranging from 3KHz to 300 MHz with a near field delivery using specialized antenna in the presence of high instantaneous magnetic field.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with clinically definite MS according to Polman
* Age 18 to 60 yrs.
* EDSS 0 to 7.
* Relapse-free > 30 days prior to inclusion.
* Stable immunomodulatory or immunosuppressive. therapy or treatment for > 3 months prior to inclusion.
* In case of treatment with antidepressants:

stable therapy > 3 months prior to inclusion.

* Highly effective methods of birth control for females.

Exclusion Criteria:

* Pregnancy
* Cardiac pacemakers, biostimulators, neurostimulators, cochlear implants, hearing aids.
* MRI incompatible implants like intramedullary nails, intracranial aneurysm clips, intra-orbital metal fragments, stents, implanted medication pumps etc near target area.
* Critically ill patients needing life support system.
* Mentally challenged patients who cannot give informed consent.
* Severely ill patients who cannot lie in supine position for 1 hour.
* H/o brain injury and/ or any malignant disorder
* Personal or family history of epilepsy / brain tumor.
* Relapse of MS < 30 days prior to inclusion
* Change of immunomodulatory therapy < 30 days prior to inclusion
* Bipolar disorder
* History of stroke or other brain lesions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Effect of RFQMR therapy on MS lesion confirmed by Magnetic Resonance Imaging (MRI) | Change from baseline to 90 days post therapy
  1. Change in number of T1 gadolinium- enhancing lesions on MRI from baseline to 90 days post therapy.
  2. Change in number of lesions on FLAIR MRI images from baseline to 90 days post therapy.
  3. Change in volume of five larger lesions of brain and spine from baseline to 90 days post therapy

SECONDARY OUTCOMES:
Effect of RFQMR therapy on disability status and quality of life of MS patients. | Change from baseline to 90 days post therapy
  1. Change in Extended Disability Status Score (EDSS) from baseline to 90 days post therapy.
  2. Change in Functional Assessment for Multiple sclerosis (FAMS) score from baseline to 90 days post therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjit Kumar, MD, Principal Investigator — SCALENE CYBERNETICS LIMITED
Locations (1):
- Centre for Advanced Research and Development, Bangalore, Karnataka, India

REFERENCES:
- [Background] Cone CD Jr. Variation of the transmembrane potential level as a basic mechanism of mitosis control. Oncology. 1970;24(6):438-70. doi: 10.1159/000224545. No abstract available. PMID 5495918